CLINICAL TRIAL: NCT00461253
Title: Case-Control-Study on the Breast Cancer Risk of Mirena® Compared With Copper IUDs
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Juergen Dinger, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2006_02
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Intrauterine Devices, Copper

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Breast Cancer Cases
  Interventions: Device: Levonorgestrel-releasing IUD; Device: Copper IUD
- 2: Matched Controls for Breast Cancer Cases
  Interventions: Device: Levonorgestrel-releasing IUD; Device: Copper IUD

INTERVENTIONS:
Device: Levonorgestrel-releasing IUD — This is a case-control-study; strictly speaking the category "intervention type" does not apply to this study.
  Other Names: Mirena
Device: Copper IUD — This is a case-control-study; strictly speaking the category "intervention type" does not apply to this study.

SUMMARY:
The objective of this study is to determine the breast cancer risk of Mirena® users compared to copper intrauterine device (IUD) users in a community-based case-control study.

DETAILED DESCRIPTION:
This is a community-based case-control study in Germany and Finland. Cases will be identified from cancer registries, tumor centers and breast centers. Matched controls will be accrued from the same region as the case came from. Breast cancer cases and their controls are women under 50 years of age without known history of malignancies.

Cases are women with a breast cancer who are younger than 50 years of age at cancer diagnosis. The breast cancer was diagnosed between January 2000 and December 2007. Only alive cases and cases in a sufficiently good health status to be interviewed are eligible for the study.

Controls are women without a breast cancer diagnosis who are younger than 50 years of age at the time of the interview. About 3 controls matched by year of birth and region will be allocated to each case.

A standardized questionnaire will be used for all breast cancer cases and controls. The questionnaire will be mailed to cases and controls.

Study participants will be asked for their informed consent. Data confidentiality according to national laws will be ensured by the field organizations.

ELIGIBILITY:
Inclusion Criteria:

* cases: women with a breast cancer who are younger than 50 years of age at cancer diagnosis
* controls: women without a breast cancer diagnosis who are younger than 50 years at the time of the interview

Exclusion Criteria:

* women who are not willing to participate

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases will be identified from population-based cancer registries, tumor centers and breast centers. Matched controls will be accrued from the same region as the case came from.
Sampling Method: Non-Probability Sample
Enrollment: 25565 (Actual)
Dates: Start 2006-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Dinger, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Result] Dinger J, Bardenheuer K, Minh TD. Levonorgestrel-releasing and copper intrauterine devices and the risk of breast cancer. Contraception. 2011 Mar;83(3):211-7. doi: 10.1016/j.contraception.2010.11.009. Epub 2011 Jan 7. PMID 21310281

RESULTS

PARTICIPANT FLOW:
Groups:
- Cases: Cases were defined as women who were diagnosed with breast cancer (invasive carcinoma or carcinoma in situ) between 1/2000 and 12/2007 and aged <50 years at diagnosis.
- Controls: Controls were selected randomly from the national population registry (Finland) or via neighborhood controls by a controlled random route method (Germany).
Period: Overall Study
Arm/Group | Cases | Controls
Started | 10093 (Identified cases) | 40250 (Identified controls)
Completed | 5113 (Analyzed cases) | 20452 (Analyzed controls)
Not Completed | 4980 | 19798
Not completed — Death | 985 | 0
Not completed — Protocol Violation | 613 | 236
Not completed — no response | 2609 | 11789
Not completed — administrative | 773 | 7773

BASELINE CHARACTERISTICS:
Population: Definitions: cases were defined as women who were diagnised with breast cancer (invasive carcinoma or carcinoma in situ) between 1/2000 and 12/2007 and aged <50 years at diagnosis. Controls were selected randomly from the national population registry (Finland) or via neighborhood controls by a controlled random route method (Germany).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 5113 | 20452 | 25565
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (5.1) | 44.2 (5.1) | 44.3 (5.1)
Gender [Number; unit: participants]
  Female | 5,113 | 20,452 | 25565
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 1815 | 7260 | 9075
  Finland | 3298 | 13192 | 16490

OUTCOME MEASURES:

1. Primary Outcome: Breast Cancer Risk
Description: Breast cancer (invasive carcinoma or carcinoma in situ) in women aged <50 years at diagnosis. Cases were excluded if they had died before study start or had a history of malignancy.
Time Frame: retrospective, January 2000 to December 2007
Population: Frequency of breast cancer (in situ and invasive) in LNG-IUD users and Cu-IUD users
Measure: Number; unit: participants
Groups:
- LNG IUD: Women who currently or ever used a LNG IUDs (Mirena) at time of breast cancer diagnosis
- Cu-IUD: Women who currently or ever used a copper IUDs at time of breast cancer diagnosis
Arm/Group | LNG IUD | Cu-IUD
Number analyzed (Participants) | 5346 | 5428
participants | 1076 | 1068
Statistical Analysis 1: Comparison: LNG IUD vs Cu-IUD; In this matched case-control study, conditional logistic regression was used to investigate the relationship between a woman being a breast cancer case or a control (dichotomous dependent variable), and a set of actual or potential prognostic factors (covariates) for breast cancer (incl. the use of Mirena). Conditional logistic regression uses a maximum likelihood approach for estimating the covariates; data are stratified and the likelihoods are computed relative to each stratum; Test type: Non-Inferiority or Equivalence — Assuming a prevalence of current Mirena use among fertile women of 8% in Finland and 2% in Germany, it was estimated that 3,500 cases and 14,000 controls would be needed to exclude a 1.5-fold breast cancer risk for Mirena users compared with users of copper IUDs; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.88 to 1.12] — Breast cancer OR for ever use of LNG-IUD vs. Cu-IUD; adjusted for BMI, family history of breast cancer, age at first birth, age at menarche and physical activity (primary analysis)
Statistical Analysis 2: Comparison: LNG IUD vs Cu-IUD; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.93 to 1.17] — Breast cancer OR for ever use of LNG-IUD vs. Cu-IUD, crude
Statistical Analysis 3: Comparison: LNG IUD vs Cu-IUD; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.52 to 1.39] — Breast cancer OR for "current use" of LNG-IUD vs. Cu-IUD at time of breast cancer diagnosis; adjusted for BMI, family history of breast cancer, age at first birth, age at first menarche, physical activity (primary analysis)
Statistical Analysis 4: Comparison: LNG IUD vs Cu-IUD; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.58 to 1.41] — Breast cancer OR for "current use" of LNG-IUD vs. Cu-IUD at time of breast cancer diagnosis, crude

ADVERSE EVENTS:
Time Frame: Retrospective population based case-control study identifying breast cancer cases in the between January 2000 and December 2007 in women younger than 50 years of age at time of diagnosis.
Groups:
- LNG IUD: Users of LNG IUDs (Mirena)
- Cu-IUD: Users of copper IUDs
Arm/Group | LNG IUD | Cu-IUD
Serious Adverse Events (participants affected / at risk) | 1085/5346 | 1130/5428
Other Adverse Events (participants affected / at risk) | 0/5346 | 0/5428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LNG IUD (N=5346) | Cu-IUD (N=5428)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1085 (1085) | 1130 (1130) — Breast cancer (in situ and invasive)

LIMITATIONS AND CAVEATS:
Limitations include information-bias, which cannot be entirely eliminated in retrospective studies. However, in this study recall is likely not to be differential between cases and controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes